CLINICAL TRIAL: NCT03705910
Title: Effects of Mobilization and Perceptive Rehabilitation on Disability and Symptoms of Patients With Fibromyalgia Syndrome- A Randomised Controlled Trial
Brief Title: Effects of Mobilization and Perceptive Rehabilitation on Patients With Fibromyalgia Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University of Lefke (Other)
Responsible Party: Principal Investigator, Beraat Alptug, Master Physiotherapist, European University of Lefke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETK00-2018-0206
Record Dates: First submitted 2018-10-07; First posted 2018-10-15 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Fibromyalgia
Keywords: proprioception; manual therapies; pain; health status; posture; sleep; fatigue; depression
MeSH Terms: conditions — Fibromyalgia; Pain; Fatigue; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome measures will be performed by an experienced physiotherapist who will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Perceptive Rehabilitation (PR-group) (Active Comparator): This treatment will include small latex cones with different resistance. In each session, over one hundred cones will be placed on a rigid wooden base using elastic strips. The patient will be asked to lie down supine on the material. Patients weigh will create pressure and reaction force to his/her body. Treatments will be 2 times a week till 8 weeks.
  The therapist will ask the patient firstly to breathe normally and feel the pressure. The patient will then perform breathing exercises and active exercises (including stretching, warming up, and cooling down) under supervision. During the session, the therapist will ask about the pressure of the cones and will correct the patient's posture.
  Interventions: Other: Perceptive Rehabilitation
- Mobilisation Techniques (Mob-group) (Active Comparator): A certified physiotherapist will perform mobilisation techniques. All participants in this group will receive treatment protocol according to the list on below. Treatments will be 2 times a week till 8 weeks.
  For this treatment, the participant should lie on a bed and change their position according to the technique (supine, position or side-lying). Also, the therapist will be changing her position according to the technique. All technique will be on the range of motion limit. For releasing techniques the therapist will apply three-dimensional pressures till 3-5 minutes, with the feeling of relaxing therapist will change the limit for the next point.
  Interventions: Other: Mobilisation Techniques
- Control Group (C-group) (No Intervention): This group will not receive any intervention during this period. C-group will attend assessments.

INTERVENTIONS:
Other: Perceptive Rehabilitation — In each session, over one hundred cones will be placed on a rigid wooden base using elastic strips. The patient will be asked to lie down supine on the material. Patients weigh will create pressure and reaction force to his/her body. Treatments will be 2 times a week till 8 weeks.
  The therapist will ask the patient firstly to breathe normally and feel the pressure. The patient will then perform breathing exercises and active exercises (including stretching, warming up, and cooling down) under supervision. During the session, the therapist will ask about the pressure of the cones and will correct the patient's posture. At the end of each session, the therapist will photograph the patient's back with the aim of documenting the pressure and hyperaemic areas.
  Arms: Perceptive Rehabilitation (PR-group)
Other: Mobilisation Techniques — A certified physiotherapist will perform mobilisation techniques. All participants in this group will receive treatment protocol according to the list on below. Treatments will be 2 times a week till 8 weeks.
  For this treatment, the participant should lie on a bed and change their position according to the technique (supine, position or side-lying). Also, the therapist will be changing her position according to the technique. All technique will be on the range of motion limit. For releasing techniques the therapist will apply three-dimensional pressures till 3-5 minutes, with the feeling of relaxing therapist will change the limit for the next point.
  Arms: Mobilisation Techniques (Mob-group)

SUMMARY:
The aim of our study is to determine and compare the effects of perceptive rehabilitation against other mobilization techniques on the treatment of fibromyalgia symptoms and disability. Participants in this study will be randomly assigned to three separate groups using a random allocation software program, the three groups receiving either perceptive rehabilitation (PR-group), mobilization techniques (Mob-group), or neither (the control group, C-group).

DETAILED DESCRIPTION:
Fibromyalgia is considered to be a chronic, widespread musculoskeletal pain syndrome. Its most common symptoms are fatigue, anxiety, depression, and lack of concentration. These symptoms may lead to a decrease in the amount of physical activity that a sufferer can accomplish. Neck and back pain will also increase as the sedentary behaviour becomes the norm (Talotta et al., 2017). The best overall way of managing fibromyalgia is still under discussion, but according to the literature, symptoms are best managed by physiotherapy (García, Nicolás, and Hernández, 2016). Different programs can also be tailored to individual fibromyalgia sufferers with the aim of reducing pain (e.g. heat agents, electrotherapy, postural exercises, aerobic exercise, aqua-therapy and manual treatment).

However, according to Bronfort et al. (2010), there is insufficient evidence supporting the effectiveness of manual therapy as a treatment for fibromyalgia. According to Reis et al. (2014), a single thoracic mobilization session was able to improve short-term heart-rate variability, although the pain was not affected by the intervention.

Paolucci et al. (2016) used a new rehabilitation tool to treat pain with an increased reliance on proprioception. Practically, the tool consisted of cones made from a latex material which were placed under the patient's back during treatment sessions. These cones were intended to improve tactile response and proprioception, the so-called perceptual surface. According to this study, the tool was able to decrease pain and help to improve function. However, it is important to understand the tool's effect on long-term rehabilitation and compare it with other treatment methods. The aim of our study is to determine and compare the effects of perceptive rehabilitation and mobilization techniques on disability and fibromyalgia symptoms.

Our study will include 90 participants, with 30 participants in each group. The PR-group and the Mob-group will receive treatments twice per week for eight weeks, a total of 16 sessions; there will be no intervention in the C-group. Another physiotherapist will assess each group before and after all the sessions. The study will be single blind. Follow-up assessments will be three and six months after the last session.

ELIGIBILITY:
Inclusion Criteria:

•Having a Fibromyalgia diagnosis according to Wolfe et al. (2016) criteria.

Exclusion Criteria:

* Having a diagnosis of chronic fatigue syndrome or myofascial pain syndrome,
* Using medicine other than simple analgesics,
* Vertebrobasilar insufficiency,
* Severe scoliosis or kyphoscoliosis,
* History of spine surgery,
* History of vertebral fracture,
* Rheumatic diseases,
* History of Benign or Malign tumour,
* Osteoporosis and conditions that cause osteoporosis,
* Presence of cardiovascular risk factors,
* Serious neurological problems,
* Psychiatric disorders,
* Chronic respiratory diseases,
* After upper motor neurone lesion,
* Attending regular physical activity or exercise class during the last 3 months.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Revised-Fibromyalgia Impact Questionnaire (FIQR) | change from baseline to the end of the 8 weeks, at the end of the 3-month and 6-month follow-up period
  Turkish version of FIQR will be use in this study. This questionnaire has 21 individual questions. All these questions should be answered according to the past 7 days. FIQR has divided to three sections; 'function, overall impact and symptoms'. The total FIQR score will be calculate with the sum of the three domain scores.

SECONDARY OUTCOMES:
Socio-demographic and clinical characteristics | change from baseline to the end of the 8 weeks, at the end of the 3-month and 6-month follow-up period
  Date of birth, sex, marital status, profession, education status, medical histories, medications, time period of body pain, time of the diagnosis of FMS, symptoms, when pain increases, which activities increases pain and complaints will be noted.
Body Mass Index (BMI) | change from baseline to the end of the 8 weeks, at the end of the 3-month and 6-month follow-up period
  Weight and height will be combined to report BMI in kg/m^2.
Postural assessment 1 | change from baseline to the end of the 8 weeks, at the end of the 3-month and 6-month follow-up period
  New York Posture Rating Chart will be used to evaluate the posture. These evaluations will be on anterior, posterior and both lateral sides of the body. Therapist will give numerous rating for any deformities that can be seen. A score is allocated to each area according to the position: 5 points to the correct position; 3 points for a slight deviation, and 1 point for a pronounced deviation. Total score is between 18-90 points. Higher the points better the postural alignment.
Postural assessment 2 | change from baseline to the end of the 8 weeks, at the end of the 3-month and 6-month follow-up period
  Posture Grid will be used to evaluate the posture. These evaluations will be on anterior, posterior and both lateral sides of the body. Therapist will note any deformities that can be seen.
Cervical flexibility tests | change from baseline to the end of the 8 weeks, at the end of the 3-month and 6-month follow-up period
  Cervical flexibility will be assessed in flexion, extension, rotation and lateral flexion according to Armiger & Martyn (2010).
Cervical joint position sense | change from baseline to the end of the 8 weeks, at the end of the 3-month and 6-month follow-up period
  The patient will have a small laser pointer mounted onto a lightweight headband, which they will wear. The patient will be seated 100 cm from the wall. Measurements will be noted on the graph paper. The starting point that is projected by the laser on the graph paper will be marked. First the patients will perform active neck movements with eyes open and than eyes closed. After movement, the patient will return their head as accurately as possible to the starting position. This will include 3 trials, which will include cervical flexion, lateral flexion. The final laser position is measured against the starting position in centimetres.
Pressure pain threshold and toleration | change from baseline to the end of the 8 weeks, at the end of the 3-month and 6-month follow-up period
  Pressure algometer will be used to assess pain threshold and toleration. Measurements will be taken from both side of the body (low cervical region, second rib, occiput, trapezius muscle and supraspinatus muscle).
Short form of McGill pain questionnaire (SF-MPQ) | change from baseline to the end of the 8 weeks, at the end of the 3-month and 6-month follow-up period
  Turkish version of Short form of McGill pain questionnaire (SF-MPQ) will be used in this study. The main section of this questionnaire includes 15 words that describe pain. Patients should mark these words according to their pain intensities on a rating scale (0:none, 1:mild, 2:moderate, 3:severe). Next section of the SF-MPQ is measurement of pain intensity according to the visual analogue scale (VAS). The last section is the evaluative total pain intensity. The total score of the main component is derived by adding the rank values given by the patient for each descriptor out of 45. Scores can range from 0 to 45. A higher score of the main component of the SF-MPQ reflects more serious pain.
Beck Depression Inventory (BDI) | change from baseline to the end of the 8 weeks, at the end of the 3-month and 6-month follow-up period
  Turkish version of Beck Depression Inventory (BDI) will be used in this study. This inventory has 21 self-report items about depressive symptoms. All items should be answered from 0 through 3. The higher score represents the more intensity of the symptom. Items should be answered according to the past 2 weeks. The total score on the BDI, which has a range of 0 to 63. Higher values represent greater severity of depression (0-9 minimal depression 10-18 mild depression 19-29 moderate depression 30-63 severe depression).
Fatigue Severity Scale (FSS) | change from baseline to the end of the 8 weeks, at the end of the 3-month and 6-month follow-up period
  Turkish version of Fatigue Severity Scale (FSS) will be used in this study. This scale has 9 items. Each item should be scored (strongly disagrees) 0 to 7 (strongly agrees). The minimum score=9 and maximum score possible=63. Higher score=greater fatigue severity. The average score for all 9 items constitutes the FSS score.
Pittsburgh Sleep Quality Index (PSQI) | change from baseline to the end of the 8 weeks, at the end of the 3-month and 6-month follow-up period
  Turkish version of Pittsburgh Sleep Quality Index (PSQI) will be used in this study. This is a self-reported index that has 19 items with Likert and open-ended response formats. This index should be answered according to the past month. Minimum Score "0" means "good sleep" and Maximum Score "21" means "disrupted sleep".

CONTACTS AND LOCATIONS:
Overall Officials: Beraat Alptug, MSc, Principal Investigator — European University of Lefke; Emine H. Tüzün, Prof. Dr., Principal Investigator — Eastern Mediterranean University; Barıs Kececi, PT, Principal Investigator — European University of Lefke; Levent Eker, M. D., Principal Investigator — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

REFERENCES:
- [Background] Bronfort G, Haas M, Evans R, Leininger B, Triano J. Effectiveness of manual therapies: the UK evidence report. Chiropr Osteopat. 2010 Feb 25;18:3. doi: 10.1186/1746-1340-18-3. PMID 20184717
- [Background] Angel Garcia D, Martinez Nicolas I, Saturno Hernandez PJ. "Clinical approach to fibromyalgia: Synthesis of Evidence-based recommendations, a systematic review". Reumatol Clin. 2016 Mar-Apr;12(2):65-71. doi: 10.1016/j.reuma.2015.06.001. Epub 2015 Oct 16. English, Spanish. PMID 26481494
- [Background] Paolucci T, Baldari C, Di Franco M, Didona D, Reis V, Vetrano M, Iosa M, Trifoglio D, Zangrando F, Spadini E, Saraceni VM, Guidetti L. A New Rehabilitation Tool in Fibromyalgia: The Effects of Perceptive Rehabilitation on Pain and Function in a Clinical Randomized Controlled Trial. Evid Based Complement Alternat Med. 2016;2016:7574589. doi: 10.1155/2016/7574589. Epub 2016 Jan 13. PMID 26884794
- [Background] Reis MS, Durigan JL, Arena R, Rossi BR, Mendes RG, Borghi-Silva A. Effects of posteroanterior thoracic mobilization on heart rate variability and pain in women with fibromyalgia. Rehabil Res Pract. 2014;2014:898763. doi: 10.1155/2014/898763. Epub 2014 May 29. PMID 24991436
- [Background] Talotta R, Bazzichi L, Di Franco M, Casale R, Batticciotto A, Gerardi MC, Sarzi-Puttini P. One year in review 2017: fibromyalgia. Clin Exp Rheumatol. 2017 May-Jun;35 Suppl 105(3):6-12. Epub 2017 Jun 28. PMID 28681712
- [Derived] Alptug B, Tuzun EH, Kececi B, Eker L. Effects of perceptive rehabilitation and mobilization methods on symptoms and disability in patients with fibromyalgia: A preliminary randomized control trial. Ir J Med Sci. 2023 Dec;192(6):2937-2947. doi: 10.1007/s11845-023-03333-6. Epub 2023 Mar 10. PMID 36897535
- See also: Armiger, P., & Martyn, M. A. (2010). Stretching for functional flexibility: Wolters Kluwer Health/Lippincott, Williams, & Wilkins. — https://books.google.com.cy/books?id=ZqlfAAAACAAJ&dq=Armiger,+P.,+%26+Martyn,+M.+A.+(2010).+Stretching+for+functional+flexibility:+Wolters+Kluwer+Health/Lippincott,+Williams,+%26+Wilkins.&hl=en&sa=X&ved=0ahUKEwihspCn6uXdAhXKkCwKHdVrA9AQ6AEILTAB